CLINICAL TRIAL: NCT00350545
Title: A Phase 2 Trial of Rituximab and Corticosteroid Therapy for Newly Diagnosed Chronic Graft Versus Host Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sally Arai, Associate Professor of Medicine (Blood and Marrow Transplantation), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-04948; 96950 (Other: Stanford University alternate IRB Number); BMT177 (Other: OnCore); NCI-2011-00450 (Other: National Cancer Institute (NCI))
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Rituximab; Prednisone; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab + prednisone arm (Experimental): Rituximab will be given as an IV fusion as initial treatment, followed by predisone (given during registration) which will be continued through-out trial and tapered off by physician. Cyclosporine A and tacrolimus will be used if chances of new diagnosis of chronic GVHD occur. Both drugs have no interaction with Rituxan, but will be tapered off after predisone is completely tapered.
  Interventions: Drug: Rituximab; Drug: Prednisone; Drug: Cyclosporine A; Drug: tacrolimus

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2;IV infusion once weekly for four doses (days 1,8,15,22); option for second 4-week course at week 9
  Other Names: Rituxan
Drug: Prednisone — 1 mg/kg; po per day with taper
  Other Names: Deltasone; Liquid Pred; Meticorten; Orasone
Drug: Cyclosporine A — trough 200-300 or lower; po
  Other Names: cyclosporine; Ciclosporin
Drug: tacrolimus — trough 5-10 or lower; po
  Other Names: FK-506; Fujimycin

SUMMARY:
The addition of rituximab to prednisone for the initial treatment of chronic GVHD will increase the overall response rate, enable a more rapid and effective steroid taper.

DETAILED DESCRIPTION:
To determine the efficacy of Rituximab as first line of treatment of chronic GVHD. Efficacy will be defined as he ability to taper prednisone to a dose of 0.25 mg/kg per day by 6 months without clinical or GVHD relapse/ recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults with a new diagnosis of chronic GVHD- that requires systemic immunosuppressive treatment to a dose of 1mg/kg/day prednisone and who have undergone any type of donor hematopoietic cell graft or conditioning regimen.
* Stable doses of other immunosuppressive medications (e.g. calcineurin inhibitors, mycophenolate mofetil) for 2 weeks prior to enrollment. In addition, these other immunosuppressive medications should not be dose increased.
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* All subjects must provide written informed consent.

Exclusion Criteria:

* Known life-threatening hypersensitivity to Rituximab or other anti-B cell antibody.
* Treatment with prednisone (or equivalent) at doses higher than 1 mg/kg/day at the time of enrollment. Persistent prednisone treatment of acute GVHD that is less than 1mg/kg is allowed.
* Active, uncontrolled infection- CMV reactivation is excluded (i.e. pneumonitis, colitis). Peripheral blood CMV reactivation is allowed as long as it is not associated with CMV disease and is responding to therapy.
* Known Hepatitis B surface Ag positive
* Active malignant disease relapse.
* Pregnancy
* Lactating
* Inability to comply with the Rituximab treatment regimen.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-08; Primary Completion 2012-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miklos, Principal Investigator — Stanford University; Sally Arai, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available in the publication which is forthcoming.

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Prednisone Arm: To determine the efficacy of Rituximab as first line of treatment of chronic GVHD.
Period: Overall Study
Arm/Group | Rituximab + Prednisone Arm
Started | 37
Completed | 35
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + Prednisone Arm
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Ability to Successfully Taper Prednisone to a Dose Lower Dose.
Description: Participants that have successfully tapered prednisone to a dose of 0.25 mg/kg/Day by 6 Months without clinical relapse.
Time Frame: 6 months
Population: Participants who have complete or partial clinical response to therapy as well as a steroid dose, tapered to <0.25 mg/kg/day within 6 months after initiation of rituximab
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Prednisone Arm
Number analyzed (Participants) | 35
Participants | 14

2. Secondary Outcome: Number of Participants With Complete and/or Partial GVHD Response
Description: To have physician documentation of clinical GVHD response using organ staging and scoring scale- NIH clinical GVHD consensus response criteria applied 6 months after rituximab infusion began
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Prednisone Arm
Number analyzed (Participants) | 35
Participants
  Complete response | 12
  Partial response | 15

3. Secondary Outcome: Participants Who Reduced Steroid Use at One Year After Enrollment on the Trial
Description: Participants that decreased total daily corticosteroids ≤ 0.25mg/kg one year after rituximab infusion began
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Prednisone Arm
Number analyzed (Participants) | 35
Participants | 14

4. Secondary Outcome: Failure-free Survival at 6 and 12 Months Post-Rituximab Initiation
Description: Failure-free survival (FFS) was defined as participants who are surviving with no relapse and second line of cGVHD treatment.
Time Frame: 6 and 12 Months
Population: At initiation of therapy, all patients were on high dose of steroids (1mg/kg/day). Failure-free survival (FFS) rate for the 31 patients at 6 and 12 months post-rituximab initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Prednisone Arm
Number analyzed (Participants) | 35
Participants
  6 month FFS | 28
  12 month FFS | 21

5. Secondary Outcome: Overall Survival
Description: Overall survival at 6 and 12 months
Time Frame: 6 and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Prednisone Arm
Number analyzed (Participants) | 35
Participants
  6 month overall survival | 33
  12 month overall survival | 30

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Rituximab + Prednisone Arm
Serious Adverse Events (participants affected / at risk) | 35/35
Other Adverse Events (participants affected / at risk) | 26/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Prednisone Arm (N=35)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6
Nocardia infection (Respiratory, thoracic and mediastinal disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 3 — on leg, fore-arm and lower extremities. Includes superficial
Abscess (Blood and lymphatic system disorders) | 3 — Including: Incision, drainage, right paraspinous muscle
Low absolute neutrophil count (Blood and lymphatic system disorders) | 1
Bacterial infection (Infections and infestations) | 1 — Including: fungal
bilirubin levels increasing (Blood and lymphatic system disorders) | 1
Blood (Blood and lymphatic system disorders) | 2 — Large amounts of blood seen in ET tube and trachea
Cardiac arrest (Cardiac disorders) | 1 — Inlcudes pulseless electrical activity
Chest pain (Cardiac disorders) | 2
Graft versus host disease (General disorders) | 12 — Including: of the- mouth, liver, skin lung and chronic
Confusion (General disorders) | 1 — (worsening)
Conjunctivitis (Eye disorders) | 1 — ( viral )
Cough (Respiratory, thoracic and mediastinal disorders) | 3 — Includes: severe and prodcutive
Death (General disorders) | 5
Diarrhea (Renal and urinary disorders) | 1 — (bloody)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Includes: worsening
Erythematous rash (Skin and subcutaneous tissue disorders) | 1 — Includes: Dry and flaky
Fever (General disorders) | 2
H1N1 (Respiratory, thoracic and mediastinal disorders) | 1
Tachycardia (Cardiac disorders) | 2
Veno-occlusive disease (Renal and urinary disorders) | 1
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1
Tbili (Renal and urinary disorders) | 2
Syncope (Blood and lymphatic system disorders) | 2
Stroke (General disorders) | 2
Sespis (Infections and infestations) | 2
Respiratory syncytial virus (Respiratory, thoracic and mediastinal disorders) | 2
Multi-organ system failure (General disorders) | 1
Ischemia (Blood and lymphatic system disorders) | 1
Disseminated aspergillus (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3 — inlcudes Isolated events
Sinus bradycardia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Prednisone Arm (N=35)
Fever (General disorders) | 3
Cellulitis (Skin and subcutaneous tissue disorders) | 1 — Includes: Superficial
Cold symptoms (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Decrease in diffusing capacity of the lungs for carbon monoxide (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pain (Gastrointestinal disorders) | 3 — Includes: pain in abdomin, on forearm,
Infections (Infections and infestations) | 2 — Includes: E.Coli
Erythematous (Skin and subcutaneous tissue disorders) | 2
Hypertensive (Blood and lymphatic system disorders) | 1
influenza A (Immune system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Orthostatic hypotension (Blood and lymphatic system disorders) | 1
Paranasal sinus disease (Respiratory, thoracic and mediastinal disorders) | 1
slight decrease in her forced expiratory volume in 1 second (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes